CLINICAL TRIAL: NCT03503630
Title: Short-course Radiation Followed by mFOLFOX-6 Plus COMPOUND 2055269 for Locally-advanced Rectal Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ali Shamseddine (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Phoenix Clinical Research (Other)
Responsible Party: Sponsor-Investigator, Ali Shamseddine, Principal Investigator, American University of Beirut Medical Center
Organization: American University of Beirut Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2017-0422; MS100070_0021 ISS (Other Grant/Funding Number: Merck KGaA, Darmstadt, Germany)
Record Dates: First submitted 2018-03-29; First posted 2018-04-20 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: Locally advanced rectal cancer; Immunotherapy; Short course radiation; Folfox; Response rate
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Locally advanced rectal cancer patients (Experimental): 1. Week 1: D1-5: radiotherapy 25 Gy in 5 fractions
  2. mFOLFOX-6: Oxaliplatin 85 mg/m2 in a 2-hour infusion Leucovorin 400 mg/m² over 2 hours Bolus fluorouracil 400 mg/m² followed by a 48-hour infusion of fluorouracil 2,400 mg/m² + COMPOUND 2055269 10 mg/kg every 2 weeks (first administration at D15, for a total of 6 cycles)
  3. Week 16 or 17 (2 to 3 weeks after last cycle of chemotherapy + COMPOUND 2055269): Total Mesorectal Excision
  Interventions: Drug: COMPOUND 2055269; Radiation: Radiation Therapy; Drug: mFOLFOX; Procedure: Total Mesorectal Excision

INTERVENTIONS:
Drug: COMPOUND 2055269 — COMPOUND 2055269 to be given every 2 weeks with chemotherapy for 6 cycles
Radiation: Radiation Therapy — Radiotherapy 25 Gy to be given on Days 1-5
Drug: mFOLFOX — Given every 2 weeks for 6 cycles
Procedure: Total Mesorectal Excision — Surgery to be done 2-3 weeks after last cycle of chemotherapy and COMPOUND 2055269

SUMMARY:
The purpose of this study is to show that the addition of COMPOUND 2055269, an immunotherapeutic drug, to Folfox chemotherapy will improve the pathologic complete response rate in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
The purpose of this study is to show that the addition of COMPOUND 2055269, an immunotherapeutic drug, to Folfox chemotherapy will improve the pathologic complete response rate in patients with locally advanced rectal cancer.

COMPOUND 2055269 has demonstrated meaningful clinical activity across various tumor types and treatment settings. No clinical trial is conducted over COMPOUND 2055269 in locally-advanced rectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years.
2. Locally-advanced rectal cancer (cT2 N1-3, cT3 N0-3, evidence of extramural vascular or mesorectal fascia involvement).
3. <12 cm from anal verge.
4. Histologically proven rectal adenocarcinoma.
5. ECOG performance score ≤ 1.
6. Have adequate organ function by meeting the following:

   * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
   * Platelet count ≥ 100 × 109/L;
   * Hemoglobin ≥ 9 g/dL;
   * Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range;
   * AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver);
   * Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft- Gault formula (or local institutional standard method).
7. Negative serum or urine pregnancy test at screening for women of childbearing potential.
8. Highly effective contraception for both male and female subjects throughout the study and for at least 30 days after last COMPOUND 2055269 treatment administration if the risk of conception exists.

Exclusion Criteria:

1. Distant metastasis (M1).
2. Patients with T2 N0 or T4.
3. Recurrent rectal cancer.
4. Symptoms or history of peripheral neuropathy.
5. Prior radiotherapy or chemotherapy.
6. Current use of immunosuppressive medication, except for the following:

   * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intraarticular injection);
   * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
   * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
7. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
8. Vaccination within 4 weeks of the first dose of COMPOUND 2055269 and while on trials is prohibited except for administration of inactivated vaccines.
9. Active infection requiring systemic therapy.
10. Known history of testing positive for the human immunodeficiency virus or known acquired immunodeficiency syndrome.
11. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
12. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
13. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
14. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
15. Prior organ transplantation including allogenic stem-cell transplantation.
16. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
17. Concurrent treatment with a non-permitted drug.
18. Patients suspected by the physician that he/she will not compliant to the protocol conduct.
19. Pregnant or breastfeeding patients.
20. Patient participating in another clinical trial.
21. Patient who is not willing to sign the consent form.
22. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
23. Legal incapacity or limited legal capacity patients receiving other oncology specific medication not authorized in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2024-07-02 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the pathologic complete response (pCR) rate following short-course radiation then mFOLFOX-6/COMPOUND 2055269 | After 17 weeks (once surgery is done)
  Will be done via pathologic assessment on the surgical specimen

SECONDARY OUTCOMES:
The proportion of patients who remain progression free at 3 years. | 3 years
  1) Progression free survival is measured by imaging and serial tumor markers during follow up visits
PD-L1 expression and T-cell infiltration changes after treatment | At day 10 biopsy and after 17 weeks (once surgery is done)
  2) PD-L1 & T cell infiltration is measured by a pathology assessment on day 10 and after surgery
Number of participants with treatment- related adverse events as assessed by NCI-CTCAE v4.0 | 3 years
  Treatment- related adverse events are assessed by NCI-CTCAE v4.0 in each visit
Quality of life of the patients in a neoadjuvant setting with COMPOUND 2055269 as assessed by FACT-C questionnaire | 3 years
  Quality of life is measured via FACT-C questionnaire in each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ali I Shamseddine, M.D., Principal Investigator — American University of Beirut Medical Center
Locations (3):
- King Hussein Cancer Center, Amman, Jordan
- Lebanon (2):
  - American University of Beirut Medical Center, Beirut
  - Hôtel Dieu de France, Beirut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shamseddine A, Zeidan YH, El Husseini Z, Kreidieh M, Al Darazi M, Turfa R, Kattan J, Khalifeh I, Mukherji D, Temraz S, Alqasem K, Amarin R, Al Awabdeh T, Deeba S, Jamali F, Mohamad I, Elkhaldi M, Daoud F, Al Masri M, Dabous A, Hushki A, Jaber O, Charafeddine M, Geara F. Efficacy and safety-in analysis of short-course radiation followed by mFOLFOX-6 plus avelumab for locally advanced rectal adenocarcinoma. Radiat Oncol. 2020 Oct 7;15(1):233. doi: 10.1186/s13014-020-01673-6. PMID 33028346
- [Derived] Shamseddine A, Zeidan YH, Kreidieh M, Khalifeh I, Turfa R, Kattan J, Mukherji D, Temraz S, Alqasem K, Amarin R, Al Awabdeh T, Deeba S, Jamali F, Mohamad I, Elkhaldi M, Daoud F, Al Masri M, Dabous A, Hushki A, Jaber O, Khoury C, El Husseini Z, Charafeddine M, Al Darazi M, Geara F. Short-course radiation followed by mFOLFOX-6 plus avelumab for locally-advanced rectal adenocarcinoma. BMC Cancer. 2020 Sep 1;20(1):831. doi: 10.1186/s12885-020-07333-y. PMID 32873251